CLINICAL TRIAL: NCT00429260
Title: A 1-week, Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of Abrupt Discontinuation of Saredutant in Outpatients With Depression Who Completed 8 Weeks of Treatment With Saredutant 100 mg Once Daily
Brief Title: A Study Evaluating the Safety and Tolerability of Abrupt Discontinuation of Saredutant in Patients With Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SFY6577; SR48968
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Depressive Disorder
Keywords: depression; antidepressive agents
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — SR 48968

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Saredutant

SUMMARY:
The primary objective is to evaluate the safety and tolerability of abrupt discontinuation of saredutant over 1 week in outpatients with depression who completed 8 weeks of treatment with saredutant 100 mg once daily.

The secondary objective is to evaluate the safety and tolerability of 8 weeks of open-label treatment with saredutant 100 mg once daily in outpatients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder,single or recurrent episode, as defined by Diagnostic and Statistical Manual of Mental Disorders DSM-IV criteria

Exclusion Criteria:

* Total score of <22 on the Montgomery-Asberg Depression Rating Scale (MADRS).
* Duration of the current depressive episode is less than 1 month or greater than 2 years.
* Total score of <25 on the Mini Mental State Examination (elderly patients ≥65 years only).
* Patients with a history or presence of bipolar disorders or psychotic disorders.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 6 months except nicotine or caffeine dependence.
* Patients who have used the following prior to entry: benzodiazepines or sedative-hypnotics more than 2 days per week within 1 month, antipsychotics within 1 month, fluoxetine within 1 month, monoamine oxidase inhibitors within 2 weeks, other antidepressants, anxiolytics, or mood-stabilizer (lithium, anticonvulsants) within 1 week.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline (Day 56) to Day 63 in the post-baseline average daily number of discontinuation-emergent signs or symptoms from the 17-item Discontinuation-Emergent Signs and Symptoms checklist.

SECONDARY OUTCOMES:
The main secondary endpoints are the change from baseline in the maximum number of post-baseline discontinuation-emergent signs or symptoms and the proportions of patients with any newly-occurring post-baseline discontinuation-emergent signs and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Administrative Office, Malvern, Pennsylvania, United States